CLINICAL TRIAL: NCT04549116
Title: A Multicenter, Randomized, Controlled, Double-blind, Double-dummy Study to Evaluate the Safety and Efficacy of Subcutaneous Progesterone Compared to Vaginal Progesterone for Luteal Phase Supplementation in Modified Natural Frozen Euploid Blastocyst Transfer.
Brief Title: Subcutaneous Progesterone in Frozen- Thawed Single Euploid Blastocyst Transfer.
Acronym: PROGRESS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20US-Prg03
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Infertility
Keywords: Frozen embryo transfer
MeSH Terms: conditions — Infertility | interventions — Crinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, double-dummy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational (Experimental): Progesterone-IBSA 25mg, twice daily (BID) subcutaneous (SC) injection every 12 hours and Crinone Placebo, once daily (QD) intravaginally.
  Interventions: Drug: Progesterone-IBSA Injectable Solution; Drug: Placebo Vaginal gel with applicator
- Comparator (Active Comparator): Crinone 8%, 90 mg, QD intravaginally and Progesterone-IBSA Placebo, BID SC Injection every 12 hours
  Interventions: Drug: Progesterone Vaginal Gel with Applicator; Drug: Placebo injectable solution

INTERVENTIONS:
Drug: Progesterone-IBSA Injectable Solution — Progesterone-IBSA 25mg, twice daily (BID) SC Injection every 12 hours
  Other Names: Prolutex
  Arms: Investigational
Drug: Progesterone Vaginal Gel with Applicator — Crinone 8%, 90 mg, QD intravaginally
  Other Names: Crinone
  Arms: Comparator
Drug: Placebo Vaginal gel with applicator — Vaginal gel Placebo, once daily (QD) intravaginally
  Arms: Investigational
Drug: Placebo injectable solution — Placebo injectable solution, BID SC Injection every 12 hours
  Arms: Comparator

SUMMARY:
This is a multicenter, randomized, double-blind, double-dummy, active-controlled, non-inferiority clinical study in women aged 35 to 42 years. This study will investigate the safety and efficacy of Progesterone-IBSA to support euploid embryo blastocyst implantation and early pregnancy after frozen embryo transfer (FET) in a modified natural cycle as a treatment for infertile women. Subjects will be randomized to receive either active Progesterone-IBSA or Crinone 8% for luteal and early pregnancy support and these two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* subject has given written informed consent;
* Premenopausal women 35 to 42 years of age at the time of consent (at least 35 [including day of birthday] and no more than 42 [up to the day before their 43rd birthday]);
* Valid indication for IVF treatment (i.e. history of infertility according to ASRM definition, single women or same-sex couples);
* Consistent, regular spontaneous ovulatory menstrual cycle with normal length (24-38 days included);
* Body mass index (BMI) < 38 kg/m2;
* Subject with at least one euploid frozen blastocyst from a previous IVF treatment cycle;
* Less than 3 previous consecutive euploid blastocyst transfers without a life birth;
* Baseline Follicle Stimulating Hormone (FSH) < 15 mIU/mL, and Anti Muellerian Hormone (AMH) >0.7 ng/mL (within 6 months from screening for subjects requiring a stimulation cycle to obtain a euploid embryo); and Estradiol (E2) < 90 pg/mL and Progesterone (P4)< 1.5 ng/mL at Visit 1 (for all subjects);
* Semen used during IVF(for subjects requiring a stimulation cycle to obtain a euploid embryo) was produced by ejaculation (not surgically derived sperm) from either the partner or from a sperm donor. Donor must be 18-40 years of age at the time of collection and compliant with 21 Code of Regulations (CFR) section 1271 Subpart C;
* Hysterosalpingography, hysteroscopy, 3D ultrasound or sonohysterogram documenting a normal uterine cavity within the last year;
* Normal cervical cytology/High Risk human papillomavirus (HPV) testing per American College of Obstetricians and Gynecologists guidelines.

Exclusion Criteria:

* Oligo or anovulation (spontaneous menses > 39 days apart);
* Breastfeeding or Pregnancy;
* Contraindication to pregnancy (i.e. an active, uncontrolled clinically significant medical condition or abnormality of the sexual organs determined by the provider);
* Known family history of major congenital anomalies;
* Moderate to severe current endometriosis (stage 3 or 4);
* Presence of a unilateral or bilateral hydrosalpinx that communicates with the uterus, that has not been ligated prior to treatment;
* Recurrent pregnancy loss (RPL) as defined by the American Society of Reproductive Medicine (ASRM) as two or more consecutive failed clinical pregnancies;
* Presence of a submucosal or intramural fibroid > 4 cm which distorts the uterine cavity or are > 5 cm in diameter;
* Untreated uterine pathology that could impair embryo implantation (i.e. scarring/Asherman's syndrome or intra uterine polyps > 1 cm in size);
* Type 1 or 2 diabetes mellitus based on American Diabetes Association (ADA) criteria3;
* Uncontrolled adrenal or thyroid dysfunction;
* History of conditions (i.e. toxic shock syndrome) that would contraindicate use of a vaginal progesterone product;
* Subjects with hepatic impairment (liver function tests > 2x upper limit of normal);
* Subjects with renal impairment (estimated creatinine clearance <60 mL/min/1.73 m2);
* History of an active or treated autoimmune disease (i.e. systemic lupus erythematosus);
* History of arterial disease (i.e. Prior or active thrombophlebitis, thromboembolic disorder or known thrombophilia);
* Neoplasias (current) or history of neoplasia that may be responsive to progesterone;
* High grade cervical dysplasia;
* Undiagnosed vaginal bleeding (i.e. at the time of screening);
* Use of donor eggs or plans to use a gestational carrier;
* Use of endometrial receptivity array (ERA) test to postpone or anticipate the embryo transfer (ET) day;
* Use of epididymal, testicular , electro-ejaculated or chemotherapy exposed sperm;
* Known allergy to progesterone preparations or their excipients;
* Current dependence on alcohol, tobacco (must not be smoking/using tobacco x 2 months before the study) or drugs or psychotropic medications labeled as Pregnancy Categories D and X;
* Use of concomitant medications within 1 month previous the start of the FET cycle preparation up to gestational week 12 that might interfere with the study evaluation (use of insulin sensitizing agents, vaginal medications/preparations, any drugs for luteal support other than those specified in the protocol, aspirin, any hormonal treatment, with the exception of levothyroxine);
* Participation in a concurrent clinical trial or in another investigational drug trial within the past 2 months-

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 680 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 5 weeks post-embryo transfer
  defined by the presence of an intrauterine fetal heart beat
Ongoing pregnancy | 10 weeks post-embryo transfer
  defined by the presence of an ongoing intrauterine pregnancy with fetal heart beat

SECONDARY OUTCOMES:
Positive pregnancy rate | 10+/-2 days after embryo transfer.
  positive serum β-human chorionic gonadotropin (hCG) test rate
Implantation rate | 6 weeks after embryo transfer,
  defined by the number of gestational sacs observed at Visit 6 by means of a transvaginal ultrasound (TVUS), divided by the number of blastocysts transferred (%)
Delivery rate | 2-4 weeks post expected delivery date.
  defined as the number of deliveries with at least one live birth or stillbirth (%)
Live birth rate | 2-4 weeks post expected delivery date.
  defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life
Cycle cancellation rate (with reason) | from treatment start until 10 weeks of pregnancy
  defined as number of subjects dropping form the study at any time.
Adverse Events related to the mother | from Informed consent signature until 2-4 week after delivery.
  frequency and severity of adverse events related to the mother.
Local tolerability | from the 4th day of treatment administration until 10 weeks post embryo transfer.
  At each visit, the subject will be queried about the presence of local reactions at administration site (pain, redness, swelling and itching at injection site and pain, irritation, swelling and leakage in the genital area). Events will be described in term of nature, severity (mild, moderate, severe, or very severe) and duration (persisted for up to 1 hour, persisted for more than 1 up to 4 hours, persisted for more than 4 up to 12 hours, persisted for more than 12 hours).
Early Miscarriage rate | from 5 weeks post embryo transfer until the 12th week of pregnancy.
  defined as a spontaneous loss of an intra-uterine pregnancy
Late miscarriage rate | after the 12th week of pregnancy until delivery.
  defined as a spontaneous loss of an intra-uterine pregnancy
Ectopic pregnancy rate | from 5 weeks post embryo transfer until the 12th week of pregnancy.
  defined as a pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology.
Adverse events related to the newborn. | 2-4 weeks after expected delivery.
  frequency and severity of adverse events related to the newborn.

OTHER OUTCOMES:
Progesterone Pharmacokinetic (PK) characterization | 4 days after treatment start.
  Blood sampling to assess Progesterone levels will be collected in order to characterize the PK profile at steady state in the target population

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - The Fertility Treatment Center, LLC, Tempe, Arizona
  - HRC Fertility, Encino, California
  - Kindbody, Los Angeles, California
  - San Diego Fertility, San Diego, California
  - Spring Fertility, San Francisco, California
  - Illume Fertility, Norwalk, Connecticut
  - Reproductive Associates of Delaware, Newark, Delaware
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - IVF Florida Reproductive Associates, Margate, Florida
  - The IVF Center, Winter Park, Florida
  - InVia Fertility Specialists, PLLP, Hoffman Estates, Illinois
  - Johns Hopkins Fertility Center, Lutherville, Maryland
  - University Reproductive Associates, PC, Hasbrouck Heights, New Jersey
  - Reproductive Endocrinology Associates of Charlotte, Charlotte, North Carolina
  - Carolina Conceptions, Raleigh, North Carolina
  - Institute for Reproductive Health, Cincinnati, Ohio
  - Main Line Fertility, Bryn Mawr, Pennsylvania
  - Shady Grove Fertility, Chesterbrook, Pennsylvania
  - Care Fertility, Bedford, Texas
  - Aspire Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, LLC., Shady Grove Fertility, Webster, Texas
  - Utah Fertility Center, PC, Pleasant Grove, Utah